CLINICAL TRIAL: NCT00051194
Title: A 6-week Safety and Efficacy Study of Combination IOP-lowering Therapy in Patients With Open-angle Glaucoma or Ocular Hypertension.
Brief Title: A 6-week Safety & Efficacy Study of Combination Intraocular Pressure-lowering Therapy in Patients With Open-angle Glaucoma or Ocular Hypertension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C-02-03
Record Dates: First submitted 2003-01-03; First posted 2003-01-07 (Estimated); Last update posted 2012-04-16 (Estimated); Status verified 2006-03

CONDITIONS: Glaucoma, Open-angle; Ocular Hypertension
Keywords: Glaucoma; POAG; OAG; OHT
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension; Glaucoma

INTERVENTIONS:
Drug: Combination IOP Lowering Therapy

SUMMARY:
To compare the intraocular pressure(IOP)-lowering efficacy of morning or evening instillations of a combination IOP-lowering therapy in patients with open-angle glaucoma or ocular hypertension.

ELIGIBILITY:
Adult patients of any race and either sex with open angle glaucoma or ocular hypertension.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-09; Primary Completion 2003-07 (Actual); Study Completion 2003-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alcon Investigators, Principal Investigator — Alcon Research
Locations (1):
- Europe, Fort Worth, Texas, United States